CLINICAL TRIAL: NCT01767220
Title: Primary Endo- and Epicardial vs. Endocardial Ablation of Sustained Ventricular Tachycardia in Patients With Underlying Cardiac Disease (VTeee)
Brief Title: Endo- and Epicardial vs. Endocardial Ablation of Ventricular Tachycardia in Patients With Cardiac Disease
Acronym: VTeee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dietmar Baensch, Prof. Dr. Dietmar Baensch, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 2012-0125
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Ventricular Tachycardia
Keywords: ventricular tachycardia; endocardial ablation; epicardial ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strategy 1- endocardial ablation (Active Comparator): VT substrate mapping and VT ablation are done only from endocardial.
  Interventions: Procedure: Strategy 1 - endocardial ablation
- Strategy 2 - endocardial and epicardial ablation (Active Comparator): VT substrate mapping and ablation are done from endocardial and epicardial.
  Interventions: Procedure: Strategy 2 - endocardial and epicardial ablation

INTERVENTIONS:
Procedure: Strategy 1 - endocardial ablation — VT substrate mapping and VT ablation are done only from endocardial. Therefore the catheters are introduced through the femoral veins/arteries. For mapping and ablation a 3,5 mm irrigated tip catheter (Navistar Thermocool, Biosense Webster, Diamond Bar, CA, USA) will be used.
  Arms: Strategy 1- endocardial ablation
Procedure: Strategy 2 - endocardial and epicardial ablation — VT substrate mapping and VT ablation are done from endocardial and epicardial. Therefore the catheters are introduced through the femoral veins/arteries and into the pericardial space via a pericardial puncture. After endocardial and epicardial mapping, ablation is done from endocardial. In case of an ineffective endocardial ablation and an epicardial substrate an epicardial ablation is done. For mapping and ablation from endo- and epicardial a 3,5 mm irrigated tip catheter (Navistar Thermocool, Biosense Webster, Diamond Bar, CA, USA) will be used.
  Arms: Strategy 2 - endocardial and epicardial ablation

SUMMARY:
A significant portion of patients with cardiac diseases like coronary artery disease (CAD), dilated cardiomyopathy (DCM) and arrhythmogenic right ventricular cardiomyopathy (ARVC) develops ventricular tachycardia (VT). The standard ablation procedure is carried out from endocardial only. In 30% of patients treated this way a successful ablation is not possible. In these cases the scar areas are mostly located in the outer layer of the myocardium. Ablation is feasible only if the catheter is placed in the epicardial space to reach the surface of the heart muscle. In the past this type of ablation was performed as a second procedure in case of recurrent VTs after unsuccessful endocardial ablation.

This prospective randomized trial compares the standard ablation procedure (endocardial ablation only) with a new strategy. This means in a single procedure the scar areas responsible for VT are marked and obliterated from endocardial as well as from epicardial. The primary endpoint is recurrence of VT after endo- and epicardial vs. endocardial ablation only.

40 patients will be enrolled. They will be randomized 1:1 in the study arms "strategy 1" which is standard endocardial ablation and "strategy 2" which is endo- and epicardial ablation.

At least 12 months are planned for enrollment. The study is closed if the patient last enrolled has completed the 12-months-follow up. Follow up visits are scheduled 3, 6 and 12 months after the ablation procedure. Recurrence of VT is monitored by ICD (implanted cardioverter defibrillator) interrogation.

Both ablation strategies are well established and conducted with standard equipment. The methodology of this study does not contain any experimental approaches. The standard insurance coverage of the hospital is guaranteed for all enrolled patients.

DETAILED DESCRIPTION:
A significant portion of patients with cardiac diseases like coronary artery disease (CAD), dilated cardiomyopathy (DCM) and arrhythmogenic right ventricular cardiomyopathy (ARVC) develops ventricular tachycardia (VT). These arrhythmia often causes symptoms like dizziness, shortness of breath, angina or even cardiogenic shock. Large trials showed that VTs are associated with a 3.4 to 5fold increase in mortality even if each episode was successfully terminated by an ICD. Initially most patients are treated with antiarrhythmics. If these drugs are ineffective or not tolerated because of side effects catheter ablation (obliteration of cardiac tissue by radiofrequency) is the only alternative therapy.

The mechanism of most VTs are reentry circuits which are typically found in areas of scar in the left or right chamber. These scar areas may be located in the inner layer of the myocardium (endocardial), in the outer layer (epicardial) or in all layers of the heart muscle (transmural). The standard ablation procedure is carried out from endocardial only. This means catheters introduced through the femoral veins or arteries are placed in the right or left ventricle. In 30% of patients treated this way a successful ablation is not possible. In these cases the scar areas are mostly located in the outer layer of the myocardium. Ablation is feasible only if the catheter is placed in the epicardial space to reach the surface of the heart muscle. In the past this type of ablation was performed as a second procedure in case of recurrent VTs after unsuccessful endocardial ablation.

This prospective randomized trial compares the standard ablation procedure (endocardial ablation only) with a new strategy. This means in a single procedure the scar areas responsible for VT are marked and obliterated from endocardial as well as from epicardial. The primary endpoint is recurrence of VT after endo- and epicardial vs. endocardial ablation only.

Patients are eligible if they show documented VT on the basis of an underlying cardiac disease and a therapy with antiarrhythmics was ineffective or not tolerated. In terms of this study cardiac disease means CAD, DCM and ARVC. All patients have to be treated with an ICD. Patients are not eligible if VT is not documented, if there is no structural heart disease, if they have a mechanical aortic valve or a pacemaker/ICD with epicardial leads implanted or if a pericardial puncture must not be done.

40 patients will be enrolled. They will be randomized 1:1 in the study arms "strategy 1" which is standard endocardial ablation and "strategy 2" which is endo- and epicardial ablation.

In case of strategy 1 ablation catheters are placed in the right, left or both ventricles through the femoral veins/arteries. VT is induced by programmed stimulation and then analysed. By means of 3D-electroanatomical mapping the endocardial surface is reconstructed. The scar areas are marked and in a second step obliterated.

In case of strategy 2 in addition to the endocardial access via femoral veins/arteries a pericardial puncture is performed to get access to the epicardial space. This allows placement of ablation catheters on the epicardial surface of the heart. VT is induced and analysed from endo- and epicardial. In addition to strategy 1 a 3D-reconstruction of the epicardial surface is made and scar areas are marked like from endocardial. In a first step endocardial ablation is performed. Thereafter changes in epicardial scar areas are analyzed. In case of still inducible VT after endocardial ablation epicardial ablation is performed as a second step. The success of strategy 1 and 2 is always checked by programmed ventricular stimulation.

At least 12 months are planned for enrollment. The study is closed if the patient last enrolled has completed the 12-months-follow up. Follow up visits are scheduled at 3, 6 and 12 months after the ablation procedure. Recurrence of VT is monitored by ICD interrogation.

Both ablation strategies are well established and conducted with standard equipment. The methodology of this study does not contain any experimental approaches. The standard insurance coverage of the hospital is guaranteed for all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* structural heart disease (CAD, DCM, ARVC)
* ICD already implanted
* documented ventricular tachycardia
* patient is able to give informed consent
* VT ablation because of vital indication

Exclusion Criteria:

* VT without structural cardiac disease
* VT not documented
* patient is not able to give informed consent
* contraindication for pericardial puncture
* mechanical aortic valve
* pacemaker or ICD with an epicardial lead

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
recurrence of any VT | up to 12 months after the date of VT ablation
  Recurrence of any VT is measured by ICD interrogation, which is routinely done at the following follow-up visits: 3, 6 and 12 months after the date of the VT ablation procedure. In case of emergency (e.g. incessant VT, VT storm, resuscitation due to ventricular fibrillation) an additional ICD interrogation is done at admission to hospital.

SECONDARY OUTCOMES:
percentage of VT substrates which can only be abolished by epicardial ablation | date of VT ablation - up to 3 to 5 days
  This secondary outcome measure is evaluated only once during the hospital stay at the date of the VT ablation procedure. The average time of hospital stay for VT ablation is estimated to 3 to 5 days.
12 lead ECG features typical for epicardial VT substrates | date of VT ablation up to 3 to 5 days
  This secondary outcome measure is evaluated only once during the hospital stay at the date of the VT ablation procedure. The average time of hospital stay for VT ablation is estimated to 3 to 5 days.
percentage of epicardial VT substrates referred to the underlying cardiac disease | date of VT ablation - up to 3 to 5 days
  This secondary outcome measure is evaluated only once during the hospital stay at the date of the VT ablation procedure. The average time of hospital stay for VT ablation is estimated to 3 to 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Baensch, Prof. Dr., Principal Investigator — University Hospital of Rostock, Dept. of Cardiology
Locations (1):
- University Hospital of Rostock, Rostock, Mecklenburg-Vorpommern, Germany